CLINICAL TRIAL: NCT00275158
Title: Effect of L-Arginine Therapy on the Glomerular Injury of Pre-Eclampsia: A Randomized Controlled Trial
Brief Title: Glomerular Injury of Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Bryan Myers, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK-52876 (completed); DK-52876
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia; Glomerular Filtration Rate (GFR); Inulin clearance; Hypertension; L-Arginine; Nitric Oxide; cGMP; Endothelin; ADMA
MeSH Terms: conditions — Pre-Eclampsia; Hypertension

INTERVENTIONS:
Drug: L-Arginine Supplementation

SUMMARY:
Pre-eclampsia complicates 7 - 10% of pregnancies and constitutes a leading cause of fetal growth retardation and premature birth, as well as infant and maternal morbidity and mortality. The kidney is the primary site of injury resulting in high blood pressure, loss of protein into the urine and decreased kidney function. The release of vasoconstrictors over vasodilators from an abnormal placenta may underlie pre-eclampsia. Nitric Oxide (NO) is an important vasodilator that is thought to play an important role in the kidneys ability to accommodate to a healthy pregnancy. Normal pregnancy in the rat is accompanied by increased production of NO and its second messenger cGMP. There is a parallel increase in renal expression of constitutive nitric oxide synthase (NOS), the enzyme that generates NO from arginine. In the pregnant rat, an infusion of NG-nitro-L-arginine methyl ester (L-NAME), an exogenous inhibitor of NOS, has been shown to replicate some of the hemodynamic features of the syndrome of pre-eclampsia. In a recent animal study, L-arginine supplementation reversed the adverse effects of L-NAME on pregnancy by attenuating the high blood pressure and by significantly decreasing protein loss in the urine. To date, studies of the use of L-arginine supplementation to treat women with pre-eclampsia have been small or uncontrolled and have only assessed blood pressure as a primary outcome measure. We report a single center, randomized, placebo-controlled trial of L-arginine supplementation for the treatment of pre-eclampsia, in which precise physiological techniques have been utilized to assess kidney dysfunction in addition to blood pressure.

DETAILED DESCRIPTION:
OBJECTIVE: To assess the benefit of L-arginine, the precursor to nitric oxide (NO), to blood pressure and recovery of the glomerular lesion in pre-eclampsia.

METHODS: 45 women with pre-eclampsia were randomized to receive either L-arginine or placebo until day 10 post-partum. Primary outcome measures including MAP, glomerular filtration rate and proteinuria were assessed on the third and tenth days postpartum by inulin clearance and albumin-to-creatinine (A/C) ratio. NO, cyclic guanosine 3'5' monophosphate (cGMP), endothelin-1 (ET) and asymmetric-dimethyl-arginine (ADMA) and arginine levels were assayed prior to delivery, on the third and tenth day postpartum. Healthy gravid women provided control values. Assuming a standard deviation of 10 mmHg, the study was powered to detect a 10 mmHg difference in MAP (alpha 0.05, beta 0.20) between the study groups.

RESULTS: No significant differences existed between the groups with pre-eclampsia prior to randomization. Compared to the gravid control group, women with pre-eclampsia did not reveal significantly depressed levels of serum arginine, but did reveal significantly increased serum levels of ET, cGMP and ADMA prior to delivery. Despite a significant increase in serum arginine levels due to treatment, no differences were found in the levels of NO, ET, cGMP or ADMA between the two groups with pre-eclampsia. Further, there were no significant differences in any of the primary outcome measures with both groups demonstrating equivalent improvements in both blood pressure and proteinuria.

CONCLUSION: Blood pressure and kidney function improve markedly in pre-eclampsia by the tenth day postpartum. L-arginine supplementation does not hasten this recovery.

ELIGIBILITY:
Inclusion Criteria:

- Women selected for the study were diagnosed with pre-eclampsia in the second half of pregnancy.

i.) an elevation of blood pressure to levels in excess of 140 systolic over 90 diastolic ii.) proteinuria determined by a urine dipstick value ≥ 2+, or quantitated at ≥ 0.5 g either per gram of creatinine or in a 24 hour urine collection.

Exclusion Criteria:

* Women with a history of underlying renal disease defined as a pre-pregnancy azotemia (serum creatinine ≥ 1.2 mg/dl) or proteinuria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2000-01; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Mean Arterial Pressure
Glomerular Filtration Rate (inulin clearance)
Proteinuria (albumin to creatinine ratio)

SECONDARY OUTCOMES:
Vasoactive hormone levels - Nitric Oxide, Endothelin, cGMP, ADMA
Neonatal Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Bryan D Myers, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States